CLINICAL TRIAL: NCT04335617
Title: A Multicenter, Randomized, Double Blind Placebo Controlled Trial of Micronized Purified Flavonoid- Fraction (MPFF) in the Management of Radiation Proctitis
Brief Title: Micronized Purified Flavonoid- Fraction (MPFF) in the Management of Radiation Proctitis
Acronym: MiFlaPRO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Collaborators: Servier Affaires Médicales (Industry)
Responsible Party: Principal Investigator, Irmgard E Kronberger, MD, Principle Investigator, Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MiFlaPRO_2019
Record Dates: First submitted 2019-12-13; First posted 2020-04-06 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Proctitis Radiation

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, double-blind, placebo-controlled Phase III study.
Who Masked: Participant, Investigator
Masking Description: In this double blinded study Daflon and placebo are packed in the same manner, the blind is also protected by randomization. Only the principal investigator can break the blind in case of ethical or threatening patterns by contacting the sponsor and clinical research item.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational (Experimental): Patients receive MMPF 500mg for one year
  Interventions: Drug: MMPF (Micronized purified Flavonoid-Fraction)
- Placebo (Placebo Comparator): Patients receive Placebo for one year
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MMPF (Micronized purified Flavonoid-Fraction) — 500mg film-coated tablet, oral route, tablets should be taken at meal times. 4-day course of 6 tablets daily, followed by 4 tablets over the next 3 days followed by 2 tablets daily, one at midday and one in the evening
  Arms: Investigational
Other: Placebo — 4-day course of 6 tablets daily, followed by 4 tablets over the next 3 days followed by 2 tablets daily
  Arms: Placebo

SUMMARY:
national and multi-center trial for medical therapy of chronic radiation proctitis inducing anorectal bleedings

DETAILED DESCRIPTION:
Radiation proctitis is an inflammation of rectal mucosa, a complication following radiation therapy for cancers of the prostate, cervix, uterus, bladder and other malignancies in the pelvic area. Around 20 % of radiation patients develop radiation proctitis. There is a significant lack of trial treatments for radiation proctitis, even more, the studies often are small and single center designed or case series. In 2 recent reviews pointing out the management of radiation proctitis (2018 and 2016) a summary of current options in therapy according to current scientific knowledge is given. Unfortunately, these studies are about interventional options with the serious risk of complication. Only little data and lack of significance in smaller series on conservative strategies are given.

The goal of the trial is to implement a specific medication in the management and every grade of radiation proctitis - concomitant to eventual need of MMPF is described with potent anti-inflammatory mucosal capacity reducing bleeding, pain and urgency symptoms in patients with hemorrhoidal and/or postoperative symptoms. By using a placebo instead of comparative oral medications (with low evidence) this study might illustrate clinical significance of expected results as well as information on the natural history of radiation proctitis.

The goal of the study is to compare the number of necessary interventions required to stop bleeding in chronic radiation proctitis in patients receiving MMPF in comparison to patients in the control group receiving Placebo within 12 months of medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent form
* male and female patients
* age ≥ 18 years
* patients with diagnosis of radiation proctitis with macroscopic bleeding
* end of radiotherapy ≥ 3 month = 90 days ago

Exclusion Criteria:

* infectious proctitis
* ulcerative proctitis (inflammatory bowel disease)
* persons unable to understand the informed consent
* persons, who are in dependent relationship with the study investigators or Sponsor
* pregnant or lactating women
* participation in an interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2023-02-26 (Estimated); Study Completion 2023-08-26 (Estimated)

PRIMARY OUTCOMES:
Number of necessary intervention | Day 1- Day 360
  Interventions to stop acute bleeding by chronic radiation proctitis: surgical, endoscopic or proctoscopic interventions

SECONDARY OUTCOMES:
Quality of life of patients | Day 0 Day 180 Day 360
  Differences in quality of life of patients will be measured with evaluation of two questionnaires (EORTC QLQ C30 & PRT20). Higher scores mean a better quality of life.
Blood samples | Day 0-Day 360
  Differences in serum hemoglobin, thrombocytes, coagulation parameters (quick/pt=prothrombin time)
Stool | Day 0-Day 360
  Differences in calprotectin stool level
Presence of histological alterations | Day 0-Day 360
  Differences in histological alterations (distortion of crypts, Inflammation of crypts, fibrosis and ectasia of vessels, cytokines)

CONTACTS AND LOCATIONS:
Locations (11):
- Austria (11):
  - Medizinische Universität Innsbruck, Innsbruck, Tyrol
  - Krankenhaus der Stadt Dornbirn, Dornbirn
  - Barmherzige Brüder Krankenhaus Graz, Graz
  - Medizinische Universität Graz, Graz
  - Universitätsklinikum Krems, Krems
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Kepleruniversität Linz, Linz
  - Universitätsklinikum Tulln, Tulln
  - Medizinische Universität Wien, Vienna
  - Krankenhaus Nord, Klinik Floridsdorf, Vienna
  - Salzkammergut Klinikum Vöcklabruck, Vöcklabruck